CLINICAL TRIAL: NCT06726395
Title: Randomized Controlled Clinical Trial Comparing Treatment With Cloxacillin Versus Benzylpenicillin in Bacteraemia Caused by Penicillin-susceptible Staphylococcus Aureus (PSSA)
Brief Title: Comparison of Cloxacillin and Benzylpenicillin in Penicillin Susceptible S. Aureus Bacteraemia
Acronym: COMeBAC
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Principal Investigator, Malin Hagstrand Aldman, PI, MD, PhD, Region Skane
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-506860-15-00; 2023-506860-15-00 (EU CTIS Number)
Record Dates: First submitted 2024-11-26; First posted 2024-12-10 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2024-11

CONDITIONS: Staphylococcus Aureus Bacteraemia; Staphylococcal Bacteraemia; Staphylococcus Aureus Bloodstream Infections (BSI; Bacteremia); Staphylococcus (S.) Aureus Infection
Keywords: Penicillin treatment; benzylpenicillin; cloxacillin; Penicillin susceptible S. aureus; Staphylococcus aureus bacteraemia
MeSH Terms: conditions — Bacteremia | interventions — Penicillin G; Cloxacillin

STUDY DESIGN:
Intervention Model Description: Observational
Masking Description: Study personal assessing the side effects, are as fara as possible unaware of what study drug is given.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Benzylpenicillin treatment (Experimental)
  Interventions: Drug: Penicillin G_1200mg
- cloxacillin (Active Comparator)
  Interventions: Drug: cloxacillin

INTERVENTIONS:
Drug: Penicillin G_1200mg — benzylpenicillin preferred dosing 1gx4
  Other Names: bensylpenicillin; benzylpenicillin
  Arms: Benzylpenicillin treatment
Drug: cloxacillin — cloxacillin 2gx4
  Arms: cloxacillin

SUMMARY:
The goal of this study is to investigate if benzylpenicillin is a better treatment option than cloxacillin in patients with penicillin-susceptible Staphylococcus aureus bacteraemia.

DETAILED DESCRIPTION:
The overall research idea of is a RCT is to test the hypothesis that benzylpenicillin is superior to cloxacillin in the treatment of PSSA bacteraemia.

Population: Adult patients (>18 years) with PSSA bacteraemia will be eligible for enrolment in the study. Exclusion criteria are allergy to penicillin, inability to give informed consent, and concomitant growth of other clinically significant bacteria in blood cultures. We are planning a nation-wide study.

Intervention: Benzylpenicillin treatment of PSSA bacteraemia will be evaluated. As soon as S. aureus has been identified in blood cultures and the susceptibility testing indicates penicillin susceptibility (Two-three days from start of treatment), patients will be randomized to continue therapy with either cloxacillin or benzylpenicillin. The duration of treatment depends on the type of infection, and details about length of therapy and dosage will be decided by the specific patient diagnosis (i.e., endocarditis, arthritis). Repeated blood cultures and echocardiography are important in the diagnostic work-up of S. aureus bacteraemia and will be included in the study protocol. Patients will also be monitored regarding adverse events, such as liver and renal impairment, rash, diarrhoea, thrombophlebitis et c., and treatment failure, relapse, and mortality.

Control: The study drug (benzylpenicillin) will be compared to cloxacillin, which is the current drug of choice for methicillin susceptible S. aureus in Sweden. Both drugs will be used at clinically recommended doses, with appropriate adjustments for renal impairment if needed. Outcome: Primary outcome is; to be alive for 90 days without any complications. Complications are defined as having any of relapse (90 days after antibiotic finished), need of change or addition of antibiotics due to side effects or treatment failure or adverse events.

ELIGIBILITY:
Inclusion Criteria:

Aged ≥18 with penicillin susceptible S. aureus bacteraemia (PSSA), and able to provide written informed consent.

Exclusion Criteria:

* allergy to penicillin,
* inability to give informed consent,
* concomitant growth of other clinically significant bacteria in blood cultures
* neutropenia

  -≥ 96h with prior antibiotics
* When the per oral follow up medication can not be flukloxacillin or penicillinV/Amoxicillin (ie prosthetic joint infection)
* Patients in terminal palliation, where death is expected within 7 days.
* Where the treating physician believes cloxacillin is not a first-line treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Survival at 90 days without any treatment complications | From enrollment to 90 days after end of treatment
  Complications are defined as having any of; relapse within 90 days after treatment finish, need of change or addition of antibiotics due to side effects or treatment failure or adverse events.

SECONDARY OUTCOMES:
Mortality at 90 days | From enrollment to 90 days after end of treatment
  All cause mortality within 90 days from enrollment
Relapse 90 days after end of treatment | From enrollment to 90 days after end of treatment
  Relapse with positive culturing from sterile sites or high suscpition of clinical relapse
Cumulative frequency of side effects within 90 days | From enrollment until 90 days.
  all side effects registered as a cumulative frequence
Cumulative frequence of change or addition of antibiotic treatment due to sideeffects or treatment failure | from enrollment to end of treatment duration up to 90 days
  Every time additional antibiotics or change in antibiotic treatment is made due to either side effects or treatment failure (according to treating doctor)
Decrease of Bacterial DNA in blood samples | From enrollment and first 5 days
  Bacterial DNA tested the first 5 days during study treatment.

OTHER OUTCOMES:
Days with intravenous antibiotics | From enrollment and until end of treatment
  Differences between treatment groups
Different outcome measures stratified by diagnosis | From enrollment and up to 90 days after end of treatment
  90 days mortality, relapse 90 days after end of treatment, cumulative side effects stratified by diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Malin Hagstrand Aldman, PhD, MD, Principal Investigator — Lund University
Locations (1):
- Skånes universitetssjukhus, Region Skåne, Lund, Sweden

IPD SHARING:
Plan to Share IPD: No
To share the IPD is not supported by the Swedish ethical comite.

REFERENCES:
- See also: CTIS — https://euclinicaltrials.eu/search-for-clinical-trials/?lang=en&EUCT=2023-506860-15-00